CLINICAL TRIAL: NCT03582475
Title: Phase Ib Trial of Pembrolizumab (MK-3475) With Platinum-Based Chemotherapy in Small Cell/Neuroendocrine Cancers of Urothelium and Prostate
Brief Title: Pembrolizumab With Combination Chemotherapy in Treating Participants With Locally Advanced or Metastatic Small Cell/Neuroendocrine Cancers of Urothelium or Prostate
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000435; NCI-2018-01120 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-06-13; First posted 2018-07-11 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Bladder Small Cell Neuroendocrine Carcinoma; Castration-Resistant Prostate Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Prostate Carcinoma Metastatic in the Bone; Prostate Neuroendocrine Neoplasm; Prostate Small Cell Carcinoma; Stage III Bladder Cancer American Joint Committee on Cancer ( AJCC) v8; Stage III Prostate Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8; Stage IVA Bladder Cancer AJCC v8; Stage IVB Bladder Cancer AJCC v8; Ureter Small Cell Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Urethral Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Etoposide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pembrolizumab, platinum-based chemotherapy) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Participants also receive standard of care chemotherapy comprising either etoposide IV on days 1-3 and cisplatin IV or carboplatin IV on day 1 (Cohort 1), or etoposide IV on days 1-3, carboplatin IV on day 1, and docetaxel IV on day 1 (Cohort 2). Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Docetaxel; Drug: Etoposide; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase Ib trial studies how well pembrolizumab works with combination chemotherapy in treating participants with small cell/neuroendocrine cancers of the urothelium or prostate that has spread to nearby tissue or lymph nodes or that has spread to other places in the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as etoposide, docetaxel, cisplatin, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab with platinum-based chemotherapy may work better in treating participants with small cell/neuroendocrine cancers of the urothelium or prostate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the preliminary efficacy of pembrolizumab (MK-3475) in combination with standard-of-care cisplatin-based chemotherapy by assessing the durable response rate (DRR), overall response rate (ORR), duration of response (DOR), and progression free survival (PFS) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and overall survival (OS) in Cohorts 1 and 2, and radiographic PFS (rPFS) by Prostate Cancer Working Group 3 (PCWG3) and prostate-specific antigen (PSA) response in Cohort 2.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of pembrolizumab in combination with etoposide and cisplatin/carboplatin or docetaxel and carboplatin assessed by parameters of adverse events (AEs).

EXPLORATORY OBJECTIVES:

I. Determine correlation of biomarkers including PD-L1 expression (PD-L1 positive >= 1% by immunohistochemistry [IHC] using 22C3 antibody), and serum and tissue molecular (including genomic, proteomic) biomarkers that may be indicative of clinic response or safety.

OUTLINE:

Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Participants also receive standard of care chemotherapy comprising either etoposide IV on days 1-3 and cisplatin IV or carboplatin IV on day 1 (Cohort 1), or etoposide IV on days 1-3, carboplatin IV on day 1, and docetaxel IV on day 1 (Cohort 2). Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days, every 9-12 weeks for up to 2 years, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of locally advanced or metastatic 1) naive small cell cancer of the bladder, urethra, or upper urinary tract, or 2) primary small cell or neuroendocrine prostate cancer will be enrolled in this study.
* Histological diagnosis of pure or mixed small cell or neuroendocrine cancer by a genitourinary pathologist is sufficient and confirmatory immunohistochemistry is not required.
* Cohort 1 will include subjects with no prior systemic chemotherapy for locally advanced or metastatic urothelial carcinoma, with the following exception(s):

  * Platinum-based chemotherapy with recurrence > 12 months from completion of therapy is permitted.
* Cohort 2 will include subjects with no prior systemic chemotherapy for primary small cell prostate cancer, with the following exception(s):

  * Platinum-based chemotherapy with recurrence > 12 months from completion of therapy is permitted.
* Cohort 2 will include subjects with prior treatments for metastatic castration-resistant prostate cancer (mCRPC) including:

  * Prior chemotherapy with 2 other agents is allowed if > 6 months elapsed from last dose (if docetaxel chemotherapy is used more than once for hormone-sensitive and for mCRPC it will be considered 1 therapy).
  * Ongoing androgen deprivation therapy with up to 2 second-generation hormonal manipulations (e.g. including but not limited to abiraterone acetate and/or enzalutamide).
  * Ongoing treatment with for bone metastasis (e.g. denosumab or zoledronic acid) is permitted.
  * Prior immunotherapy with sipuleucel-T is allowed if completed > 4 weeks prior to trial enrollment.
* A male participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of pembrolizumab or 180 days after chemotherapy and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) or
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of pembrolizumab or 180 days after chemotherapy.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated within 6 months of screening. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. In addition, the availability of fresh frozen tissue is encouraged. Newly obtained biopsies are preferred to archival tissue.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation.
* Absolute neutrophil count (ANC) >= 1500/uL within 10 days prior to the start of study treatment.
* Platelets >= 100 000/uL (microliter) within 10 days prior to the start of study treatment.
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L within 10 days prior to the start of study treatment.

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels >1.5 x institutional ULN within 10 days prior to the start of study treatment.

  * Creatinine clearance (CrCl) should be calculated per institutional standard.
* Total bilirubin =< 1.5 ?ULN or direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ? ULN within 10 days prior to the start of study treatment.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 ? ULN (=< 5 ? ULN for participants with liver metastases) within 10 days prior to the start of study treatment.
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 ? ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants within 10 days prior to the start of study treatment.

Exclusion Criteria:

* Has disease suitable for local treatment with curative intent.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to first dose of trial treatment.

  * Note: Participants must have recovered from all AEs due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible.
  * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette?Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

  * For Cohort 1, a history of prostate cancer that was identified incidentally following cystoprostatectomy for bladder cancer is acceptable provided that the PSA is < 0.2.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV).
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (bacillus tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject?s participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Chin, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Gu Y, Ly A, Rodriguez S, Zhang H, Kim J, Mao Z, Sachdeva A, Zomorodian N, Pellegrini M, Li G, Liu S, Drakaki A, Rettig MB, Chin AI. PD-1 blockade plus cisplatin-based chemotherapy in patients with small cell/neuroendocrine bladder and prostate cancers. Cell Rep Med. 2024 Nov 19;5(11):101824. doi: 10.1016/j.xcrm.2024.101824. Epub 2024 Nov 12. PMID 39536751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened for accrual with the first enrollment on January 11, 2019. The study closed to accrual on May 5, 2022.
Groups:
- Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer: Participants receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Participants also receive standard of care chemotherapy comprising etoposide IV on days 1-3 and cisplatin IV or carboplatin IV on day 1 (Cohort 1). Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Cisplatin: Given IV
  Docetaxel: Given IV
  Etoposide: Given IV
  Pembrolizumab: Given IV
- Cohort 2: Small Cell or Neuroendocrine Prostate Cancer: Participants receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Participants also receive standard of care chemotherapy comprising etoposide IV on days 1-3, carboplatin IV on day 1, and docetaxel IV on day 1 (Cohort 2). Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Treatment Period
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Started | 7 | 8
Completed | 7 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow-up Period
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Started | 7 | 8
Completed | 7 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Customized [Count of Participants; unit: Participants]
  >50<=60 years | 1 | 3 | 4
  >60<=70 years | 3 | 4 | 7
  >70<=80 years | 2 | 1 | 3
  >80 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Durable Response Rate (DRR) (Cohorts 1 and 2)
Description: Durable Response Rate (DRR) defined as the proportion of patients who achieved a confirmed complete or partial response (CR or PR) and maintained that response for at least 6 months.
Time Frame: At 6 months
Population: one patient withdrew Cohort 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
percentage of participants | 100 | 66.7

2. Primary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Cohorts 1 and 2)
Description: Overall Response Rate (ORR) defined as patients by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 exhibited a complete or partial response (CR or PR). CR defined as disappearance of all target lesions. PR defined as >= 30% decrease in sum of the longest diameter of target lesions. .
Time Frame: Up to 3 years
Population: one patient withdrew Cohort 2
Measure: Number; unit: proportion of participents
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
proportion of participents | 0.43 | 0.43

3. Primary Outcome: Duration of Response (DOR) Per RECIST 1.1 (Cohorts 1 and 2)
Description: Duration of Response (DOR) defined as the time from the first documented CR or PR until radiograph disease progression or Prostate-Specific Antigen (PSA) progression.
Time Frame: From the first documented CR or PR up to 3 years
Population: one patient withdrew Cohort 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
Months | NA [NA to NA] — Median DOR is Not Available (NA) because none of the patients with a confirmed CR or PR had experienced radiographic or PSA progression at data cutoff. Over 50% remained progression-free, so the median could not be estimated. | 12.6 [3.15 to NA] — median, upper and lower bounds of 95% Confidence Interval could not be estimated due to insufficient number of participants with events

4. Primary Outcome: Proportion of Participants With Progression Free Survival at 12 and 24 Months
Description: Progression Free Survival (PFS) defined as the time from the first day of study treatment to first documented disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 as a 20% increase in the sum of the longest diameter of target lesions, a measurable increase in a non-target lesion, or the appearance of new lesion(s).
Time Frame: 12 months and 24 months.
Population: Proportion of Participants with Progression Free Survival at 12 and 24 Months was measured using sample size of each cohort and incidence of events to provide confidence intervals.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
Proportion of patients
  12 months | 0.86 [0.63 to 1.00] | .43 [0.18 to 1.00]
  24 months | 0.86 [0.63 to 1.00] | 0.14 [0.02 to 0.88]

5. Primary Outcome: Proportion of Participants With Overall Survival of Cohort 1 and 2 at 12 and 24 Months
Description: Overall Survival (OS) defined as the time from the first day of study treatment to the time of death from any cause.
Time Frame: 12 months and 24 months.
Population: one patient withdrew Cohort 2
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
Proportion of patients
  12 months | 0.86 [0.63 to 1.00] | 0.71 [0.45 to 1.00]
  24 months | 0.86 [0.63 to 1.00] | 0.57 [0.30 to 1.00]

6. Primary Outcome: Portion of Participants With Radiographic Progression-free Survival (rPFS) by Prostate Cancer Working Group 3 (PCWG3) at 12 and 24 Months (Cohort 2)
Description: PCWG3 is specifically designed for prostate cancer and incorporates both soft tissue and bone response assessment. RECIST 1.1 is used for evaluating responses in solid tumors, while PCWG3 combines Response evaluation criteria in solid tumors (RECIST)1.1 for soft tissue assessment with specific criteria for bone scans. The PCWG3 response criteria was used to report the portion of participants with rPFS at their 12 and 24 month assessments.
Time Frame: 12 months and 24 months.
Population: The Primary outcome of Radiographic PFS (rPFS) with response criteria based off Prostate Cancer Working Group 3 (PCWG3) only applies to Prostate cancer patients enrolled into cohort 2. This criteria does not apply to Bladder cancer patients that enrolled in Cohort 1.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 0 | 7
proportion of participants
  12 Months |  | .43 [0.18 to 1.00]
  24 Months |  | 0.14 [0.02 to 0.88]

7. Primary Outcome: Percentage of Participants With Adverse Events Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (Cohorts 1 and 2)
Time Frame: Up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
percentage of participants
  Grade 3 or higher | 57 | 25
  All Grades | 100 | 75

8. Other Pre Specified Outcome: Percentage of Participants With Programmed Death-ligand 1 (PD-L1) Combined Positive Score (CPS) Greater Than 10, at 12 Months
Time Frame: at 12 months
Population: PD-L1% (defined CPS>10). combined positive score (CPS). CPS defined as number of PD-L1 staining cells in tumor, lymphocytes, and macrophages divided by total number viable tumor cells x 100.
Measure: Number; unit: Percentage of patients with (CPS) > 10
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
Number analyzed (Participants) | 7 | 7
Percentage of patients with (CPS) > 10 | 42.8 | 37.5

ADVERSE EVENTS:
Time Frame: Adverse events are collected form consent to 90 days post treatment with a median follow up of 34 months.
Arm/Group | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 3/7 | 3/8
Serious Adverse Events (participants affected / at risk) | 7/7 | 7/8
Other Adverse Events (participants affected / at risk) | 7/7 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer (N=7) | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer (N=8)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Artirial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrolyte Toxicity (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis due to urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Metastatic or Locally Advanced Naive Small Cell Bladder Cancer (N=7) | Cohort 2: Small Cell or Neuroendocrine Prostate Cancer (N=8)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 6 (12) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
B-12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Bicep tendon tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Body odor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Breast nodularity (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchial thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Covid-19 infection (Infections and infestations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (5) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 3 (3)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Edema (General disorders) | 3 (4) | 2 (3)
Electrolyte toxicity (Metabolism and nutrition disorders) | 2 (11) | 1 (3)
Elevated liver function tests (Investigations) | 1 (6) | 0 (0)
Eye disorders (Eye disorders) | 2 (2) | 1 (4)
Fatigue (General disorders) | 7 (10) | 4 (6)
Flu like symptoms (General disorders) | 4 (4) | 1 (3)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Groin pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Grover's disease (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematologic toxicity (Blood and lymphatic system disorders) | 2 (12) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoalbuminea (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Incisional pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 3 (5)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (8)
Nausea (Gastrointestinal disorders) | 6 (8) | 4 (4)
Oral Mucositis (Gastrointestinal disorders) | 2 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (8)
Rectal fullness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Shallow breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin telangiectasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (4) | 1 (3)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Weight loss (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT03582475/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT03582475/ICF_001.pdf